CLINICAL TRIAL: NCT05488301
Title: Effects of Chest Physiotherapy in Hyperventilation Syndrom : a Multicentric Observational Study
Brief Title: Effects of Chest Physiotherapy in Hyperventilation Syndrome
Acronym: SHV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier des Pays de Morlaix (Other)
Responsible Party: Principal Investigator, Marc Beaumont, Principal Investigator, Centre Hospitalier des Pays de Morlaix
Other Study IDs: CHPMorlaix; CEPRO 2021-028 (Registry Identifier: SPLF)
Record Dates: First submitted 2022-05-27; First posted 2022-08-04 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Hyperventilation
Keywords: hyperventilation; quality of life; dyspnea; Nijmegen; anxiety
MeSH Terms: conditions — Hyperventilation; Dyspnea; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: chest physiotherapy — chest physiotherapy session including:
  * nasal ventilation
  * decrease of respiratory rate without increasement of Tidal volume
  * abdomino-diaphragmatic ventilation

SUMMARY:
Hyperventilation syndrome induce dyspnea and altered quality of life. the aim of this study is to assess the impact of chest physiotherapy on hyperventilation syndrome' symptoms

ELIGIBILITY:
Inclusion Criteria:

* patients addressed for hyperventilation syndrome
* patient aged 18 years or over
* patient able to consent and having sign a consent form

Exclusion Criteria:

* respiratory disease (COPD, interstitial lung disease, bronchiectasis, cystic fibrosis, uncontrolled asthma)
* patient with an inability to complete questionaires
* refusal of participation
* patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hyperventilation syndrome adressed for chest physiotherapy
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
change of Nijmegen score | 5 weeks
  Nijmegen score is measured at baseline and after 5 weeks. The Nijmegen questionnaire allows to assess hyperventilation symptoms. the minimum and maximum values are between 0 to 64, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
change of Nijmegen Score | 1 week
  Nijemegen score is measured at baseline and after 1 week. The Nijmegen questionnaire allows to assess hyperventilation symptoms the minimum and maximum values are between 0 to 64, and higher scores mean a worse outcome.
change of Hospital Anxiety and Depression score (HAD) | 5 weeks
  Anxiety and depression scores are measured at baseline and after 5 weeks. the minimum and maximum values are between 0 to 21 for each item (Anxiety and Depression), and higher scores mean a worse outcome.
change of Short Form-36 score (SF-36) | 5 weeks
  SF 36 score is measured at baseline and after 5 weeks. SF36 allows to assess quality of life.
  the minimum and maximum values are between 0 to 100, and higher scores mean a better outcome.
change of Dyspnea-12 score | 5 weeks
  Dyspnea-12 is measured at at baseline and after 5 weeks.
  Dyspnea-12 questionnaire allows to assess sensorial and emotional component of dyspnea. The minimum and maximum values are between à to 36, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- BEAUMONT, Morlaix, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chenivesse C, Similowski T, Bautin N, Fournier C, Robin S, Wallaert B, Perez T. Severely impaired health-related quality of life in chronic hyperventilation patients: exploratory data. Respir Med. 2014 Mar;108(3):517-23. doi: 10.1016/j.rmed.2013.10.024. Epub 2013 Nov 7. PMID 24269004
- [Background] Kiesel K, Burklow M, Garner MB, Hayden J, Hermann AJ, Kingshott E, McCullough G, Ricard R, Stubblefield G, Volz J, Waskiewicz D, Englert A. EXERCISE INTERVENTION FOR INDIVIDUALS WITH DYSFUNCTIONAL BREATHING: A MATCHED CONTROLLED TRIAL. Int J Sports Phys Ther. 2020 Feb;15(1):114-125. PMID 32089963